CLINICAL TRIAL: NCT02335632
Title: Effect of Probiotics on Gut-Liver Axis of Alcoholic Hepatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, Department of Internal Medicine, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPAH
Record Dates: First submitted 2015-01-06; First posted 2015-01-12 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Alcoholic Liver Disease
Keywords: Hepatitis; Probiotics; Lipopolysaccharides; Cytokines; Alcoholics
MeSH Terms: conditions — Liver Diseases, Alcoholic; Hepatitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): For Probiotics, 7 days
  Interventions: Drug: Placebo
- Probiotics (Active Comparator): Probiotics of 120 mg/day for 7days
  Interventions: Drug: Probiotics (Lacidofil®)

INTERVENTIONS:
Drug: Probiotics (Lacidofil®) — 7 days of cultured Lactobacillus rhamnosus R0011/acidophilus R0052 (120 mg/day)
  Other Names: Lacidofil®
  Arms: Probiotics
Drug: Placebo — For probiotics
  Other Names: For probiotics
  Arms: Placebo

SUMMARY:
Background/Aims:

The investigators explored the therapeutic effects of probiotics in patients with AH.

Methods:

Between December 2012 and January 2015, the investigators conducted a 7-day, double-controlled, randomized, prospective clinical trial comparing the efficacy of probiotics in improving liver enzymes, LPS, pro-inflammatory cytokines, stool culture, and stool Polymerase chain reaction denaturing gradient gel electrophoresis. AH was defined as an aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 and elevated AST (ALT) level with an alcohol consumption history within 48 hours. Patients were randomized to receive 7 days of cultured Lactobacillus rhamnosus R0011/acidophilus R0052 (120 mg/day) or placebo. The levels of liver enzymes, modified Discriminant Function (mDF), LPS, and pro-inflammatory cytokines, stool culture, and stool Polymerase chain reaction denaturing gradient gel electrophoresis were checked at baseline and again after therapy.

DETAILED DESCRIPTION:
Background/Aims: Alcoholic hepatitis (AH) is one of the leading causes of liver diseases. Gut-derived microbial lipopolysaccharide (LPS) has been known as a central role in the pathogenesis of AH. Some animal studies suggested an emerging role of probiotics in restoration of the bowel flora and improving liver enzymes. We explored the therapeutic effects of probiotics in patients with AH.

Methods:

Between December 2012 and January 2015, the investigators conducted a 7-day, double-controlled, randomized, prospective clinical trial comparing the efficacy of probiotics in improving liver enzymes, LPS, pro-inflammatory cytokines, stool culture, and stool Polymerase chain reaction denaturing gradient gel electrophoresis. AH was defined as an aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 and elevated AST (ALT) level with an alcohol consumption history within 48 hours. Patients were randomized to receive 7 days of cultured Lactobacillus rhamnosus R0011/acidophilus R0052 (120 mg/day) or placebo. The levels of liver enzymes, modified Discriminant Function (mDF), LPS, and pro-inflammatory cytokines, stool culture, and stool Polymerase chain reaction denaturing gradient gel electrophoresis were checked at baseline and again after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic hepatitis (AST/ALT >2 & elevated AST (ALT) level
* Alcohol >60 g/day (M), >40 g/day (F) during 7 days before screening
* Last drinks: within 48 hours prior to admission)

Exclusion Criteria:

* viral hepatitis,
* autoimmune hepatitis,
* pancreatitis,
* hemochromatosis,
* Wilson's disease,
* Drug-Induced Liver Injury,
* cancer,
* infection need for antibiotics,
* severe AH, or
* obesity (BMI >30 kg/m2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
liver enzymes | 7 days after probiotics

SECONDARY OUTCOMES:
LPS and pro-inflammatory cytokines | 7 days after probiotics
Stool culture and stool Polymerase chain reaction denaturing gradient gel electrophoresis | 7 days after probiotics